CLINICAL TRIAL: NCT07152353
Title: Clinical Trial of the Safety and Efficacy of IBA Proton Therapy System PROTEUS® PLUS (Sichuan)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ion Beam Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBA-02-CD
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
Keywords: Proton Therapy
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other): Subjects will undergo radiation therapy using the investigational medical device (PROTEUS® PLUS) in accordance with the prescribed treatment plan.
  Interventions: Device: Proton Beam Therapy (PBT)

INTERVENTIONS:
Device: Proton Beam Therapy (PBT) — PROTEUS® PLUS

SUMMARY:
This trial will enroll 47 subjects who will be be treated with the IBA PROTEUS® PLUS Proton Beam radiation Therapy (PBT) medical device.

The trial aims to assess the safety and efficacy of PROTEUS® PLUS for radiation therapy to oncology patients, and to provide a clinical basis for product registration application.

DETAILED DESCRIPTION:
The trial is structured in two distinct phases. Phase 1 - Clinical Trial: This phase spans from the initial screening through to 90 days post-treatment. Its primary objective is to assess the efficacy and safety of PROTEUS® PLUS in accordance with the regulatory requirements set by the National Medical Products Administration (NMPA) for product registration. Phase 2 - Long-Term Follow-Up: Extending up to five years after treatment, this phase aims to monitor the long-term efficacy and safety of PROTEUS® PLUS. Periodic reports will be submitted in compliance with NMPA guidelines.

ELIGIBILITY:
Inclusion Criteria (main):

* Clinically diagnosed with benign/malignant intracranial tumor and malignant solid tumor of head and neck, chest, abdomen, spine, pelvic cavity and limbs
* At least 1 lesion of the tumor to be treated is measurable according to RECIST criteria
* Expected survival time of more than 6 months
* ECOG performance status of 0 to 2
* Negative pregnancy test (HCG) results within 7 days prior to the first treatment for females of childbearing potential

Exclusion Criteria (main):

* Contraindications to radiation therapy
* Presence of other uncontrolled tumors other than the tumor to be treated
* Implants and devices in the treatment area
* Re-irradiation
* Other conditions that are not suitable for inclusion, as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Short term efficacy evaluation | 90 days after the treatment completion
  Disease Control Rate (DCR) according to Response Evaluation Criteria in Solid Tumors RECIST Version 1.1 (RECIST 1.1) criteria
Short term safety evaluation | 90 days after the treatment completion
  Toxicity of grade 3, 4 and 5 according to CTCAE

SECONDARY OUTCOMES:
Additional short term Safety evaluation | 90 days after the treatment completion
  Toxicity of grade 1 and 2 according to CTCAE
Long term Efficacy evaluation | 6 months, 1 year, 2 years, and 5 years after the end of the last treatment
  Disease Control Rate (DCR)
Long term Safety evaluation | 6 months, 1 year, 2 years, and 5 years after the end of the last treatment
  Toxicity of grade 1,2, 3, 4 and 5 according to CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Lang Jinyi, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No